CLINICAL TRIAL: NCT04845958
Title: An Observational National Pediatric Study on Prevalence of Unexplained Splenomegaly
Brief Title: A Non-Interventional National Study in Pediatric Patients With Unexplained Enlarged Spleen
Acronym: OPPUS
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS16092; U1111-1267-2545 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Gaucher Disease, Splenomegaly; Acid SphingoMyelinase Deficiency
MeSH Terms: conditions — Gaucher Disease; Splenomegaly; Niemann-Pick Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric Patients with Unexplained Enlarged Spleen

SUMMARY:
Primary Objective:

To assess prevalence of Gaucher disease (GD) diagnosed in pediatric patients presenting with unexplained splenomegaly (SMG) after exclusion of first intention-diagnoses (e.g. portal hypertension, haematological malignancy, hemolytic anemia, infection) based on clinical examination and routine biological tests (full blood count, reticulocytes, liver tests, abdominal ultrasound, Coombs test and Epstein Barr virus serology).

Secondary Objectives:

* To describe the rate of each identified disease category and the rate of patients with no final diagnosis at the end of the study in pediatric patients with unexplained SMG after exclusion of first intention diagnoses
* To describe the characteristics (clinical, lab, genetics) of all pediatric patients included in the study and to describe the characteristics subdivided by identified disease category and absence of final diagnosis at the end of the study

DETAILED DESCRIPTION:
The planned duration of this study is 39 months, which includes 36 months of patient recruitment.

ELIGIBILITY:
Inclusion criteria:

* Patient under the age of 18 years
* Patient with unexplained SMG (SMG defined as a palpable spleen, already known or discovered for the first time) and who has undergone tests to eliminate obvious causes of SMG

Exclusion criteria:

Patient with any obvious cause of SMG as described by clinical examination and/or lab or imaging test available in medical records and/or having been diagnosed with any of the following conditions:

1. hemolytic anemia
2. hematological malignancy
3. portal hypertension
4. infectious disease associated with SMG (Cytomegalovirus, Epstein Barr virus, leishmaniasis or other obvious infectious cause revealed by the medical history)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient under 18 year-old with unexplained SMG (SMG defined as a palpable spleen, already known or discovered for the first time) and who has undergone tests to eliminate obvious causes of SMG including: hemolytic anemia, hematological malignancy, portal hypertension, infectious disease associated with SMG
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Percentage of patients diagnosed with GD among enrolled patients | Up to 3 months after inclusion
  Diagnosis of GD based on deficient β-glucocerebrosidase activity in peripheral blood leukocytes or other nucleated cells, or genetic analysis.

SECONDARY OUTCOMES:
Rate of each identified disease category at the end of the study among enrolled patients | Up to 3 months after inclusion
Rate of patients with no final diagnosis at the end of the study among enrolled patients | Up to 3 months after inclusion
Number of patients based on specific char. (clinical, lab, genetics) | Up to 3 months after inclusion
  Detailed characteristics of all patients included in the study (clinical, lab, genetics) will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (40):
- France (40):
  - Investigational Site Number 2500036, Amiens
  - Investigational Site Number 2500014, Angers
  - Investigational Site Number 2500034, Argenteuil
  - Investigational Site Number 2500039, Bayonne
  - Investigational Site Number 2500015, Besançon
  - Investigational Site Number 2500003, Bordeaux
  - Investigational Site Number 2500038, Brest
  - Investigational Site Number 2500026, Caen
  - Investigational Site Number 2500018, Chambéry
  - Investigational Site Number 2500009, Clermont-Ferrand
  - Investigational Site Number 2500008, Colombes
  - Investigational Site Number 2500028, Créteil
  - Investigational Site Number 2500006, Dijon
  - Investigational Site Number 2500010, Gleizé
  - Investigational Site Number 2500031, Jossigny
  - Investigational Site Number 2500040, La Rochelle
  - Investigational Site Number 2500007, La Tronche
  - Investigational Site Number 2500030, Limoges
  - Investigational Site Number 2500001, Lyon
  - Investigational Site Number 2500032, Mantes-la-Jolie
  - Investigational Site Number 2500005, Marseille
  - Investigational Site Number 2500027, Meaux
  - Investigational Site Number 2500002, Montpellier
  - Investigational Site Number 2500021, Nantes
  - Investigational Site Number 2500019, Nice
  - Investigational Site Number 2500022, Nîmes
  - Investigational Site Number 2500016, Paris
  - Investigational Site Number 2500013, Perpignan
  - Investigational Site Number 2500035, Poissy
  - Investigational Site Number 2500011, Poitiers
  - Investigational Site Number 2500029, Reims
  - Investigational Site Number 2500023, Rennes
  - Investigational Site Number 2500037, Roubaix
  - Investigational Site Number 2500024, Rouen
  - Investigational Site Number 2500017, Saint-Priest-en-Jarez
  - Investigational Site Number 2500004, Strasbourg
  - Investigational Site Number 2500033, Toulouse
  - Investigational Site Number 2500020, Tours
  - Investigational Site Number 2500025, Valenciennes
  - Investigational Site Number 2500012, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org